CLINICAL TRIAL: NCT06753500
Title: Intraoperative Autonomic Blockade to Prevent Early Postoperative Pain After Laparoscopic Cholecystectomy: A Double-Blind, Randomized Controlled Trial
Brief Title: Intraoperative Autonomic Blockade for Laparoscopic Cholecystectomy
Acronym: ANB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Simón Bolívar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-CEI-USB-CE-0394-03
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Visceral Pain; Analgesia; Opioid Use; Postoperative Nausea; Postoperative Vomiting
Keywords: autonomic neural blockade,; Visceral pain; postoperative nausea; Postoperative vomiting; analgesic consumption; opioid use
MeSH Terms: conditions — Visceral Pain; Agnosia; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: randomized, parallel assignment, Double-Blind (Participant, Investigator), Preventive
Who Masked: Participant, Investigator
Masking Description: Randomization will be conducted using sealed envelopes stratified by the institution in blocks of six. The data manager will prepare and store the randomization list, and only they will have access to it during the study. The sealed envelopes will be placed in the patient's medical record and opened only when the patient is in the operating room and general anesthesia has been initiated. Both the patient and the independent investigator evaluating the data will remain blinded to the treatment group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autonomic Neural Blockade (Experimental): This group will receive the Autonomic nerve block performed with:
  * Bupivacaine: 20 mL of 0.5%.
  * Dexamethasone: 8 mg. Procedure: Percutaneous injection under direct laparoscopic visualization into the hepatoduodenal ligament and the visceral peritoneal reflection.
  Interventions: Procedure: Autonomic neural blockade
- NO BLOCKADE (No Intervention): Patients will undergo a laparoscopic cholecystectomy without an autonomic neural blockade

INTERVENTIONS:
Procedure: Autonomic neural blockade — Autonomic nerve block performed with:
  * Bupivacaine: 20 mL of 0.5%.
  * Dexamethasone: 8 mg.
  Other Names: BLOCKADE
  Arms: Autonomic Neural Blockade

SUMMARY:
This study proposes infiltrating the hepatoduodenal ligament and the serosal reflection of the gallbladder cystic plate with a combination of Bupivacaine (a long-acting local anesthetic) and Dexamethasone (a corticosteroid). This technique aims to block the hepatic branches of the celiac plexus to improve visceral pain control and its associated clinical manifestations, reduce analgesic requirements, and lower readmission rates, thereby facilitating recovery.

DETAILED DESCRIPTION:
Introduction

Laparoscopic cholecystectomy is the second most commonly performed procedure by general surgeons. While laparoscopy results in shorter recovery times and less intense pain compared to open surgery, it does not entirely eliminate postoperative pain, which remains the primary reason for hospitalization or readmission. Consequently, most patients undergoing laparoscopic cholecystectomy require hospitalization for 24 to 48 hours.

Postoperative pain frequently occurs after cholecystectomy, stemming from surgical incisions, manipulation of surrounding tissues, and postoperative inflammation. Various methods for pain control have been investigated, including analgesics, anti-inflammatory medication, peripheral nerve blocks, and physical interventions.

This study proposes infiltrating the hepatoduodenal ligament and the serosal reflection of the gallbladder cystic plate with a combination of Bupivacaine (a long-acting local anesthetic) and Dexamethasone (a corticosteroid). This technique aims to block the hepatic branches of the celiac plexus to enhance visceral pain control and its associated clinical manifestations, reduce analgesic requirements, and lower readmission rates, thereby facilitating recovery.

Justification

To date, no studies have shown the effect of visceral blockade on postoperative pain control in laparoscopic cholecystectomy. With the advancement of minimally invasive surgery, outpatient management of patients has become a realistic goal, presenting a challenge for surgeons to achieve adequate pain control and quicker recovery. Blocking the hepatoduodenal ligament provides an alternative for managing visceral pain by targeting the hepatic branches of the celiac plexus.

Objectives

General Objective To evaluate the effect of intraoperative infiltration of Bupivacaine and Dexamethasone into the hepatoduodenal ligament and the visceral peritoneum reflection of the gallbladder cystic plate (autonomic blockade) on postoperative pain and analgesic requirements in patients undergoing laparoscopic cholecystectomy.

Specific Objectives

1. To evaluate whether autonomic blockade reduces the consumption of postoperative opioid analgesics.
2. To assess whether autonomic blockade shortens hospital stay duration.
3. To determine whether autonomic blockade decreases the incidence of nausea and vomiting during the immediate postoperative period.
4. To evaluate the impact of autonomic blockade on hospitalization requirements (versus outpatient surgery) and the rate of readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Elective or emergency laparoscopic cholecystectomy for cholelithiasis with or without cholecystitis.

Exclusion Criteria:

* Associated biliary pathologies (e.g., biliary pancreatitis, cholangitis).

  * Additional procedures, such as formal bile duct exploration. Conversion to an open approach
  * Anesthesia or Surgical complications that require intensive care unit
* Allergies to local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesic doses | up to 72 hours
  acetaminophen 1g oral tablets
postoperative analgesic doses-rescue 1 | up to 72 hours
  Ibuprofen 400 mg oral tablets
postoperative analgesic doses-rescue 2 | up to 72 hours
  acetaminophen 300 mg plus codeine 8 mg oral tablets
postoperative analgesic-rescue 3 | up to 72 hours
  Ketorolac (30 mg) + Hyoscine (20 mg) intramuscular ampules

SECONDARY OUTCOMES:
pain level | 1, 24 and 48 hours after surgery
  Visual Analog Scale (VAS) scores will be recorded (0-10)

OTHER OUTCOMES:
postoperative nausea | 1,8 and 24 hours after surgery
  presence of nausea
postoperative vomiting | 1,8,24 hours after surgery
  presence of vomiting

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Clinica Portoazul, Barranquilla, Atlantivo
  - clinica Iberoamerica, Barranquilla, Atlántico

IPD SHARING:
Plan to Share IPD: Yes
the raw data of the study( all IPD that underlie results in a publication) will be shared with the reviewers of the correspondent Journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: during the review process in the indicated Journal
Access Criteria: though the corresponding Journal"s editorial manager.

REFERENCES:
- [Result] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Result] Daes J, Pantoja R, Luquetta J, Luque E, Hanssen A, Rocha J, Morrell DJ. Impact on Anesthetic Agent Consumption After Autonomic Neural Blockade as Part of a Combined Anesthesia Protocol: A Randomized Clinical Trial. Anesth Analg. 2024 Sep 1;139(3):581-589. doi: 10.1213/ANE.0000000000006769. Epub 2023 Dec 13. PMID 38091501
- [Result] Daes J, Pauli E. Autonomic Neural Blockade in Minimally Invasive Surgery. JAMA Surg. 2024 Dec 1;159(12):1433-1434. doi: 10.1001/jamasurg.2024.2334. PMID 39382864
- [Derived] Daes J, Hanssen A, Luque E, Mercado J, De la Rosa DG, Pauli EM. Effect of intraoperative autonomic neural blockade on early postoperative outcomes after laparoscopic cholecystectomy: a double-blind randomized controlled trial. Surg Endosc. 2026 Jan 13. doi: 10.1007/s00464-025-12542-2. Online ahead of print. PMID 41530355